CLINICAL TRIAL: NCT03075345
Title: Testing the Added Benefit of Acceptance and Commitment Therapy (ACT) in the Treatment of Obesity: a Pilot Randomised Controlled Trial.
Brief Title: Acceptance and Commitment Therapy in the Treatment of Obesity: Pilot.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: NHS service understaffing which made study unable to begin.
Sponsor: University of Sheffield (Other)
Collaborators: Mid Yorkshire Teaching NHS Trust (Other)
Responsible Party: Principal Investigator, Sarah Wakefield, Trainee Clinical Psychologist, University of Sheffield
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 151261
Record Dates: First submitted 2017-03-04; First posted 2017-03-09 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Obesity, Acceptance and Commitment Therapy, Weight Management Service
MeSH Terms: conditions — Obesity | interventions — Acceptance and Commitment Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (weight management intervention) (Active Comparator): 6 session weight management programme (over 12 weeks).
  Interventions: Behavioral: Treatment as usual (dietetic intervention)
- Treatment as usual plus acceptance and commitment therapy (Experimental): 6 session weight management programme (over 12 weeks) plus a 4 session acceptance and commitment therapy (ACT) programme. The ACT part will commence straight after the conclusion of the weight management programme.
  Interventions: Behavioral: Acceptance and commitment therapy; Behavioral: Treatment as usual (dietetic intervention)

INTERVENTIONS:
Behavioral: Acceptance and commitment therapy — Four sessions of the ACT protocol will be psychoeducational in nature, with brief experiential exercises in the class and in-between session practice. It's aim is to allow individuals to be able to sit with difficult experiences (rather than fight against them) and in turn this may allow them to live towards what they value in life.
  Arms: Treatment as usual plus acceptance and commitment therapy
Behavioral: Treatment as usual (dietetic intervention) — Six sessions of a dietetic intervention will be psychoeducational in nature around weight and nutrition, delivered by professionals working in the service.

SUMMARY:
Obesity is an 'epidemic' within the UK. Individuals living with obseity are at risk of developing cancer, heart problems and dieing. Furthermore, obesity impacts on psychological wellbeing via lowered self-efficacy, self-esteem, body image and overall quality of life (QoL). A pilot randomised controlled trial (RCT) is proposed to investigate the additional benefit of a psychological intervention alongside treatment as usual (TAU) in a weight management service. Patients routinely attending an outpatient clinic will be randomised into TAU with or without additional acceptance and commitment Therapy (ACT) group based-input and their outcomes monitored over time.

DETAILED DESCRIPTION:
Overweight and obesity is reported as an 'epidemic' problem within the UK as well as the world. Individuals living with this may be at higher risk of developing co-morbidities, such as cancers, heart problems or diabetes, and higher mortality rates are reported in this group. Furthermore, overweight and obesity can also impact on a person's psychological wellbeing, such as their self-efficacy, self-esteem and body image as well as have a negative effect on their overall quality of life (QoL). Therefore, a pilot randomised controlled trial (RCT) is proposed to investigate the additional benefit of a psychological intervention alongside treatment as usual (TAU) in a weight management service. Patients routinely attending an outpatient clinic will be randomised into TAU with or without additional Acceptance and Commitment Therapy (ACT) group based-input.

ELIGIBILITY:
Inclusion Criteria:

* Individuals will be willing and able to give informed consent for participation in the study;
* Male or Female, aged 18 years or above.
* Individuals will have a Body Mass Index (BMI) of over 40 (or over 35 if they are from a black or other minority ethic (BME) group or have a co-existing physical health problem);
* Individuals will be on a waiting list for a weight loss management programme in the UK;
* Individuals will have English as a written language.

Exclusion Criteria:

* Individuals who are currently pregnant or breastfeeding;
* Individuals with current drug or alcohol abuse, such that would prevent them from engaging in a weight management programme;
* Individuals who are acutely mentally unwell, such that would prevent them from engaging in a weight management programme;
* Individuals who at time of referral are at significant risk to themselves of others, such that would prevent them from engaging in a weight management programme;
* Individuals who are acutely physically unwell and/or hospitalised, such that would prevent them from engaging in a weight management programme;
* Individuals who have a learning disability or cognitive impairment, such that would prevent them from engaging in a weight management programme.
* Currently in receipt of psychiatric services.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05 (Estimated); Primary Completion 2017-10 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | 7 days
  A measure of psychological distress in relation to anxiety and depression symptoms. There is a total of 14 items (7 items relate to anxiety; 7 items relate to depression) with answers scored on a Likert scale of 0-3 (scores from 0-42; higher scores indicating worse symptoms).

SECONDARY OUTCOMES:
Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) | 24 hours
  The SF-36 is a generic measure of health related quality of life. There is a total of 36 questions which can be grouped into 3 levels: i) 36 individual items; ii) 8 subscales; iii) 2 summary measures.
Eating Self-Efficacy Scale (ESES) | 24 hours
  It measures self-efficacy. It contains 25-items measuring the person's confidence in ability to manage overeating in various situations (Likert scale 1-7 used).
Action and Acceptance Questionnaire - II (AAQ-II) | 24 hours
  The AAQ-II is a measure of experiential avoidance (i.e., attempts to alter difficult internal experiences which often leads to increased distress) and psychological inflexibility. Patients are asked to rate their experiences on a 7-point Likert scale (from '1: never true' to '7: always true').

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sheffield, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No